CLINICAL TRIAL: NCT06253884
Title: A Prospective Pilot Study to Evaluate the Safety, Tolerability and Technical Feasibility of Utilizing Carbon Dioxide (CO2) for Assessing Coronary Blood Flow in Subjects With Coronary Artery Disease
Brief Title: Utilizing Carbon Dioxide for Assessing Coronary Blood Flow in Subjects With Coronary Artery Disease
Acronym: NIMO-CAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12319
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Coronary Artery Disease (CAD) Subjects (Experimental): Subjects with a of coronary artery disease will undergo computer-controlled gas challenges.
  Interventions: Device: RespirAct

INTERVENTIONS:
Device: RespirAct — RespirAct device-based computer-controlled gas delivery at different concentrations as per protocol

SUMMARY:
This is a prospective pilot study to evaluate the safety, tolerability and technical feasibility of utilizing carbon dioxide for assessing coronary blood flow in subjects with coronary artery disease.

DETAILED DESCRIPTION:
The purpose of this study is to noninvasively assess changes in the heart's blood flow through inducing changes in the amount of carbon dioxide in the participant's blood and having them breathe various combinations of carbon dioxide and oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > 18 years of age
2. Clinically stable individuals with suspected or known coronary artery disease (CAD)
3. The SPECT/PET study indicates at least a mild to moderate myocardial ischemia (>5-9%) or fractional-flow-reserve (FFR) of <0.75.

Exclusion Criteria:

1. Prior myocardial infarction by clinical history (subjects with prior coronary revascularization without myocardial infarction will not be excluded)
2. Hypotension (systolic blood pressure < 100 mmHg)
3. Significant non-coronary cardiac disease (e.g., valvular abnormality, or cardiomyopathy, etc.)
4. Inability to schedule the research study within 30 days of the SPECT/PET study and prior to any coronary revascularization procedure
5. Inability to voluntarily increase their breathing rate if prompted to do so
6. Persons with mechanically, magnetically, or electrically activated implants (such as cardiac pacemakers, neurostimulators, and infusion pumps), with ferromagnetic implants or foreign bodies (such as intracranial, aneurysm clips, shrapnel, and intraocular metal chips)
7. Persons who are pregnant, nursing, or implanted with intrauterine devices (IUD's)
8. Persons with a history of significant heart, lung, kidney, or liver disease
9. Persons with asthma
10. Persons who have abnormal cardiac rhythm and rate
11. Persons unable to tolerate MRI secondary to an inability to lie supine for 60-90 minutes or severe claustrophobia
12. Persons whose renal function test does not meet MRI contrast protocol requirements [estimated Glomerular filtration rate (eGFR) < 40 mL/min/1.73m2]
13. Persons with a known history of allergy to gadolinium-based contrast
14. Enrollment in another research study.
15. Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Ratio of Maximum Signal Intensity (MSI) by BOLD MRI | 3 hours
  Maximum Signal Intensity (MSI) quantification will be measured through myocardial perfusion by blood oxygen level dependent (BOLD) MRI. The ratio of MSI in hypercarbia vs normocarbia will be evaluated in the 17-segment LV model.
Ratio of Maximum Signal Intensity (MSI) by FFP MRI | 3 hours
  Maximum Signal Intensity (MSI) quantification will be measured through myocardial perfusion by first pass perfusion (FFP) MRI. The ratio of MSI in hypercarbia vs normocarbia will be evaluated in the 17-segment LV model.

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No